CLINICAL TRIAL: NCT03982017
Title: Heart Failure Self-care Mobile Application to Reduce Readmissions Trial
Acronym: HF-SMART
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient enrollment was initially suspended due to COVID19 pandemic, then the study was closed due to institutional requirements for clinical trials.
Sponsor: University of Pittsburgh (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amber Johnson, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY18110012; K12HS019461 (AHRQ)
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Heart Failure
Keywords: readmission; quality of life; self-care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Consists of routine care at the time of hospital discharge, to be provided at the discretion of the clinicians caring for the participant.
  Interventions: Other: Usual care
- Application (Experimental): Participants will be provided a special link to navigate to the online content and resources.
  Interventions: Other: Mobile Health Technology Platform

INTERVENTIONS:
Other: Mobile Health Technology Platform — When the participant navigates to the program, s/he will follow the directions on how to use the program, sign the terms of agreement, put in a password and begin the welcome page. The participant will receive daily prompts to complete brief questionnaires and review specialized content.
  Other Names: Smartphone Program
  Arms: Application
Other: Usual care — Routine care at the time of hospital discharge, to be provided at the discretion of the clinicians caring for the participant.
  Arms: Usual care

SUMMARY:
This is a patient-centered comparative effectiveness feasibility pilot designed to examine an intervention to increase heart failure self-care and symptom recognition. The investigators will randomize 100 participants to receive either usual care at the time of discharge after heart failure admission or a smartphone application that enhances self-care.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient admission for acute decompensated heart failure
* Left ventricular systolic or diastolic heart failure
* Owns a smartphone with a data plan

Exclusion Criteria:

* Hospice or life expectancy less than 6 months
* Palliative inotrope use
* Heart transplant listed, or status post transplant
* Ventricular assist devise present, or awaiting placement
* Not being discharged to home
* Unable to provide consent or comply with the intervention
* Current enrollment in a remote monitoring/ telehealth program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Percent of participants readmitted within 30 days | 30 days post index discharge
  30-day readmission rate as determined by participant report or medical record query
Percent of participants readmitted within 90 days | 90 days post index discharge
  90-day readmission rate as determined by participant report or medical record query
Time to readmission | from the date of enrollment until the date of first documented admission or date of death from any cause, whichever comes first, assessed up to 90 days
  time to readmission
Kansas City Cardiomyopathy Questionnaire at 30 days post enrollment | 30 days post index discharge
  Quality of life, subjective level of function
Kansas City Cardiomyopathy Questionnaire at 90 days post enrollment | 90 days post index discharge
  Quality of life, subjective level of function

CONTACTS AND LOCATIONS:
Overall Officials: Amber E Johnson, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnson AE, Routh S, Taylor CN, Leopold M, Beatty K, McNamara DM, Davis EM. Developing and Implementing an mHealth Heart Failure Self-care Program to Reduce Readmissions: Randomized Controlled Trial. JMIR Cardio. 2022 Mar 21;6(1):e33286. doi: 10.2196/33286. PMID 35311679